CLINICAL TRIAL: NCT06678204
Title: Enhancing Self-care Strategies in Radiation Therapy Patients Through Diverse Smart and Flipped Education Compared to Traditional Text Booklets
Brief Title: Evaluating Illustrated Vs. Traditional Pamphlets for Enhancing Self-Care in Radiation Therapy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-A-037; 2024-A-037 (Other Grant/Funding Number: Chung Shan Medical University)
Record Dates: First submitted 2024-10-29; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-08

CONDITIONS: Radiation Therapy; Head Neck Cancer; Breast Cancer Invasive
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Optimized illustrated pamphlets (Experimental): Participants in the experimental group received optimized illustrated educational pamphlets designed to enhance understanding of self-care during radiation therapy (RT). These pamphlets included images with key text highlights tailored for better cognitive retention. Pretests were administered before the start of treatment, and posttests were conducted two weeks after the completion of RT.
  Interventions: Other: Optimized illustrated pamphlets

INTERVENTIONS:
Other: Optimized illustrated pamphlets — Participants in the control group received traditional text-based pamphlets covering similar self-care information for RT. Pretests were administered before the start of treatment, and posttests were conducted two weeks after the completion of RT.

SUMMARY:
This quasi-experimental study utilized a pre- and post-test design with experimental and control groups to assess the effectiveness of optimized illustrated educational pamphlets in enhancing patient self-care cognition, satisfaction, and reducing anxiety. The experimental group received pamphlets with a combination of images and highlighted text, while the control group received traditional text-based pamphlets. The study targeted patients undergoing radiation therapy (RT) for head and neck or breast cancer for the first time. Pre-tests assessed baseline self-care cognition, and post-tests were conducted two weeks after treatment completion. The primary objective was to improve patient awareness and understanding of self-care, aiming to support both mental and physical well-being during RT.

DETAILED DESCRIPTION:
This quasi-experimental, pre- and post-test comparison study was conducted from November 2, 2023, to August 31, 2024, at a medical center in Central Taiwan, following Institutional Review Board approval (IRB No. CS2-23058). A total of 200 first-time RT patients with head and neck or breast cancer were enrolled and randomized into two groups of 100 patients each. The experimental group received optimized illustrated pamphlets covering essential RT information, common side effects, and self-care principles, while the control group received traditional text-based pamphlets.

ELIGIBILITY:
Inclusion Criteria:

* participants with clear consciousness.
* participants could understand and comprehend Mandarin Chinese.

Exclusion Criteria:

* participants with impaired consciousness or decreased cognitive abilities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-11-02 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Self-Care Cognition | Pre-test administered before treatment and post-test two weeks after treatment completion.
  Description: Assesses patients' knowledge of radiation therapy self-care, including treatment regimen, side effects, and principles.
  Tool: Self-Care Knowledge Questionnaire (SCKQ), scored on a 0-10 scale. Higher scores indicate greater self-care knowledge.
Satisfaction with Educational Materials | Post-test administered two weeks after treatment completion.
  Description: Measures patient satisfaction with the educational materials (illustrated vs. text), with a focus on clarity and usefulness.
  Tool: Patient Satisfaction Scale (PSS), scored on a 0-5 scale. Higher scores indicate greater satisfaction.
Anxiety Assessment | Pre-test administered before treatment and post-test two weeks after treatment completion.
  Description: Evaluates patient anxiety related to radiation therapy, using the Hamilton Anxiety Rating Scale (HAMA).
  Tool: Hamilton Anxiety Rating Scale (HAMA), scored on a 0-56 scale. Higher scores indicate higher anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No